CLINICAL TRIAL: NCT02879084
Title: Variations in Retinal Nerve Fiber Layer Thickness During Uncomplicated Anterior and Intermediate Uveitis
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-3170
Record Dates: First submitted 2016-08-04; First posted 2016-08-25 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anterior Uveitis; Intermediate Uveitis
MeSH Terms: conditions — Uveitis, Anterior; Uveitis, Intermediate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates the variations in the retinal nerve fiber layer (RNFL) thickness during uncomplicated anterior and intermediate uveitis, respectively. The objectives are to 1 ) confirm the RNFL thickening during an uncomplicated anterior uveitis as described in the literature, 2) measure the RNFL thickness during an uncomplicated intermediate uveitis specifically and 3) describe the variation in time of RNFL thickness during the two types of uveitis.

DETAILED DESCRIPTION:
Thirty six individuals (18 with anterior uveitis and 18 with intermediate uveitis) will be recruited at the Centre universitaire d'ophtalmologie du CHU de Québec. RNFL thickness will be measured with optical coherence tomography at 3 times. For anterior uveitis, the RNFL thickness will be measured at presentation, 1 week and 4 to 6 weeks. For intermediate uveitis, the RNFL thickness will be measured at presentation, 4 to 6 weeks and 4 months. The initial thickness will be studied for each type of uveitis and progression over time will be studied also for each type of uveitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* anterior uncomplicated uveitis or intermediate uncomplicated uveitis

Exclusion Criteria:

* history of uveitis in the past, other than the actual uveitis
* history of ophthalmologic pathology with potential impact on retinal nerve fiber layer thickness
* optic nerve or macular clinically apparent edema
* history of glaucoma or other optic neuropathy
* suspected or confirmed multiple sclerosis
* ocular hypertension (intraocular pressure more than 22 mmHg)
* reduced optical coherence tomography signal (lower than 7) on the Cirrus HD-OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult of 18 years old or more with anterior or intermediate uncomplicated uveitis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer Thickness in anterior uveitis | At time 0
Retinal Nerve Fiber Layer Thickness in intermediate uveitis | At time 0
Change from Baseline Retinal Nerve Fiber Layer Thickness in anterior uveitis | at 4 to 6 weeks
Change from Baseline Retinal Nerve Fiber Layer Thickness in intermediate uveitis | at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon Couture, Doctor, Principal Investigator — Centre de recherche du CHU de Québec : Université Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement. CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No